CLINICAL TRIAL: NCT00784693
Title: A PHASE 2, 16 WEEK, MULTICENTER, RANDOMIZED, DOUBLE BLIND PLACEBO CONTROLLED, PARALLEL GROUP PROOF OF CONCEPT STUDY EVALUATING THE EFFICACY AND SAFETY OF TANEZUMAB FOR THE TREATMENT OF PAIN ASSOCIATED WITH ENDOMETRIOSIS
Brief Title: A Clinical Study To Investigate The Effectiveness And Safety Of Tanezumab In Treating Pain Associated With Endometriosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Further recruitment into the study was ceased on 10th December 2009, not attributed to safety. All patients recruited in the study completed all study visits.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091023; ENDOMETRIOSIS POC (Other: Alias Study Number)
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; pain; tanezumab; nerve growth factor; questionnaires
MeSH Terms: conditions — Endometriosis; Pain; Hereditary Sensory and Autonomic Neuropathies | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tanezumab (Experimental)
  Interventions: Biological: Tanezumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Tanezumab — 15 mg IV single dose
  Arms: Tanezumab
Drug: Placebo — Placebo IV single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether tanezumab is effective and safe in the treatment of pain associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menstrual women with moderate to severe endometriosis. The diagnosis of endometriosis must have been confirmed surgically within the last 8 years.
* Subjects should have regular menstrual cycle (21 - 35 days) and must be willing to use adequate contraception (2 forms of birth control, one of which must be a barrier method). Contraception is required throughout the study (screening to 16 weeks post treatment), even if subjects discontinue prematurely.

Exclusion Criteria:

* Previous hysterectomy
* Surgical treatment for endometriosis within last 6 months.
* Medical treatment for endometriosis other than combined oral contraceptive pill within the last 3 months
* Current use of the coil or progesterone only contraceptive (the combined oral contraceptive pill is allowed).
* Any history of malignant disease (cancer)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2010-01-27 (Actual); Study Completion 2010-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Bay Area Physicians for Women, Mobile, Alabama
  - Springhill Medical Center, Mobile, Alabama
  - Wilmax Clinical Research, Mobile, Alabama
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Nature Coast Clinical Research, LLC, Crystal River, Florida
  - Jacksonville Center for Clnical Research, Jacksonville, Florida
  - Advanced Women's Healthcare, West Palm Beach, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Radiant Research, Overland Park, Kansas
  - Women's Healthcare Group, Overland Park, Kansas
  - N.E.C.C.R, Fall River LLC, Fall River, Massachusetts
  - Beyer Research - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Lyndhurst Clinical Research, Kernersville, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Planned Parenthood of Arkansas and Eastern Oklahoma, Tulsa, Oklahoma
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Greenville Hospital System University Medical Group, Department of OB/GYN, Greenville, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Whitaker's Women Care, East Ridge, Tennessee
  - Advances In Health, Inc., Houston, Texas
  - Allon Health Care, Houston, Texas
  - Old Farm Obstetrics and Gynecology, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Women's Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091023&StudyName=A%20Clinical%20Study%20To%20Investigate%20The%20Effectiveness%20And%20Safety%20Of%20Tanezumab%20In%20Treating%20Pain%20Associated%20With%20Endometriosis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab: A single dose of tanezumab (RN624 or PF-04383119) 15 milligram (mg) intravenous infusion on Day 1. Participants were followed up to Week 16.
- Placebo: A single dose of placebo matched to tanezumab intravenous infusion on Day 1. Participants were followed up to Week 16.
Period: Overall Study
Arm/Group | Tanezumab | Placebo
Started | 23 | 25
Treated | 22 | 25
Completed | 20 | 19
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Randomized but not Treated | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication and completed greater than or equal to (>=)12 days of baseline observation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab | Placebo | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.7) | 30.4 (6.4) | 30.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Endometriosis Pain Score at Week 8
Description: Participants assessed daily endometriosis pain on an 11-point Numeric Rating Scale (NRS) of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores over 28 days in the baseline observation period. Post-baseline value was calculated as mean of the scores over the 28-day period preceding the post-baseline visit.
Time Frame: Baseline, Week 8
Population: Restricted full analysis set (rFAS) included all randomized participants who received at least 1 dose of study medication and completed >=12 days of baseline observation period and who had provided baseline and primary efficacy data for >=12 days of the baseline and >=15 days of each of first 2 post-randomization 28-day observation periods.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Baseline | 5.45 (1.218) | 5.50 (1.363)
  Change at Week 8 | -2.88 (2.653) | -3.51 (1.714)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 8: Analysis was based on analysis of co-variance (ANCOVA) model with main effects of treatment, contraceptive use and baseline severity of pain; Test type: Superiority or Other; Least Squares Mean Difference = 0.41, 90% CI 2-sided [-0.87 to 1.69], Standard Error of Mean 0.75

2. Secondary Outcome: Average Daily Endometriosis Pain Score at Weeks 4, 12, and 16
Description: Participants assessed daily endometriosis pain on an 11-point NRS of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores over 28 days in the baseline observation period. Post-baseline value was calculated as mean of the scores over the 28-day period preceding the post-baseline visit.
Time Frame: Weeks 4, 12, and 16
Population: Restricted FAS. Here 'number analyzed' signifies those participants who were evaluable at specified time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Week 4 | 3.55 (1.999) | 2.94 (1.814)
  Week 12: number analyzed (Participants) | 14 | 14
  Week 12 | 2.22 (2.113) | 1.45 (1.631)
  Week 16: number analyzed (Participants) | 12 | 12
  Week 16 | 3.12 (2.320) | 2.15 (2.338)

3. Secondary Outcome: Average Daily Endometriosis Pain Score During Menstruation at Baseline, Weeks 4, 8, 12, and 16
Description: Endometriosis pain during menstruation was derived from the average endometriosis pain severity as recorded on an 11-point NRS of 0 to 10 (0 = no pain and 10 = pain as bad as you can imagine) over the episode of menstruation (at least 3 days of spotting or bleeding) for the 28-day period in baseline observation period and preceding each post-baseline visit. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: Restricted FAS. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline | 6.04 (1.377) | 6.54 (1.756)
  Week 4 | 3.98 (2.503) | 3.72 (2.155)
  Week 8: number analyzed (Participants) | 17 | 13
  Week 8 | 2.99 (2.724) | 2.18 (1.540)
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | 2.92 (2.801) | 1.52 (2.117)
  Week 16: number analyzed (Participants) | 9 | 12
  Week 16 | 4.66 (2.297) | 2.94 (2.847)

4. Secondary Outcome: Average Daily Non-Menstrual Endometriosis Pain Score at Baseline, Weeks 4, 8, 12, and 16
Description: Non-menstrual endometriosis pain was derived from the average endometriosis pain severity as recorded on an 11-point NRS of 0 to 10 (0 = no pain and 10 = pain as bad as you can imagine) on the non-menstrual days for the 28-day period in baseline observation period and preceding each post-baseline visit. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Baseline | 5.25 (1.617) | 5.21 (1.348)
  Week 4 | 3.42 (1.935) | 2.77 (1.885)
  Week 8 | 2.38 (2.240) | 1.81 (2.038)
  Week 12: number analyzed (Participants) | 14 | 14
  Week 12 | 1.98 (2.124) | 1.33 (1.513)
  Week 16: number analyzed (Participants) | 12 | 12
  Week 16 | 2.86 (2.341) | 1.91 (2.288)

5. Secondary Outcome: Worst Daily Endometriosis Pain Score at Baseline, Weeks 4, 8, 12, and 16
Description: Participants assessed worst endometriosis pain in the last 24 hours on an 11-point NRS of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores over 28 days in the baseline observation period. Post-baseline value was calculated as mean of the scores over the 28-day period preceding the post-baseline visit.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Baseline | 6.20 (1.265) | 6.84 (1.297)
  Week 4 | 4.21 (2.053) | 4.00 (2.216)
  Week 8 | 3.20 (2.465) | 2.64 (2.373)
  Week 12: number analyzed (Participants) | 14 | 14
  Week 12 | 3.02 (2.612) | 2.18 (2.465)
  Week 16: number analyzed (Participants) | 12 | 12
  Week 16 | 3.87 (2.477) | 3.12 (2.818)

6. Secondary Outcome: Worst Daily Endometriosis Pain Score During Menstruation at Baseline, Weeks 4, 8, 12, and 16
Description: Participants assessed worst endometriosis pain during menstruation in the last 24 hours on an 11-point NRS of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores over the episode of menstruation (at least 3 days of spotting or bleeding) for the 28-day period in the baseline observation period. Post-baseline value was calculated as mean of the scores over the episode of menstruation (at least 3 days of spotting or bleeding) for the 28-day period preceding the post-baseline visit.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline | 6.98 (1.084) | 7.67 (1.632)
  Week 4 | 4.78 (2.532) | 5.02 (2.488)
  Week 8: number analyzed (Participants) | 17 | 13
  Week 8 | 3.60 (3.022) | 3.19 (2.356)
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | 3.58 (3.198) | 2.34 (3.072)
  Week 16: number analyzed (Participants) | 9 | 12
  Week 16 | 5.54 (2.752) | 4.03 (3.306)

7. Secondary Outcome: Worst Daily Non-Menstrual Endometriosis Pain Score at Baseline, Weeks 4, 8, 12, and 16
Description: Participants assessed worst endometriosis non-menstrual pain in the last 24 hours on an 11-point NRS of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores on non-menstrual days for the 28-day period in the baseline observation period. Post-baseline value was calculated as mean of the scores on non-menstrual days for the 28-day period preceding the post-baseline visit.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Baseline | 5.86 (1.629) | 6.60 (1.299)
  Week 4 | 4.06 (2.038) | 3.75 (2.360)
  Week 8 | 2.99 (2.331) | 2.37 (2.527)
  Week 12: number analyzed (Participants) | 14 | 14
  Week 12 | 2.79 (2.646) | 2.03 (2.358)
  Week 16: number analyzed (Participants) | 12 | 12
  Week 16 | 3.61 (2.475) | 2.85 (2.807)

8. Secondary Outcome: Average Pain Score With Intercourse at Baseline, Weeks 4, 8, 12, and 16
Description: Pain related to sexual intercourse was defined as the discomfort or pain that may occur during or after sexual intercourse with vaginal penetration. Participants assessed pain during or after sexual intercourse on an 11-point NRS of 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Higher score indicated greater pain. Baseline value was calculated as mean of the scores over 28 days in the baseline observation period. Post-baseline value was calculated as mean of the scores over the 28-day period preceding the post-baseline visit.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Baseline | 5.21 (3.209) | 5.19 (2.757)
  Week 4: number analyzed (Participants) | 13 | 12
  Week 4 | 3.32 (2.687) | 3.03 (2.298)
  Week 8: number analyzed (Participants) | 12 | 13
  Week 8 | 2.70 (2.884) | 2.92 (2.869)
  Week 12: number analyzed (Participants) | 13 | 9
  Week 12 | 2.99 (2.485) | 2.57 (2.337)
  Week 16: number analyzed (Participants) | 10 | 11
  Week 16 | 3.29 (2.976) | 3.05 (2.442)

9. Secondary Outcome: Endometriosis Symptom Severity Score (ESSS) Total Score at Baseline, Weeks 4, 8, 12, and 16
Description: Investigator assessed the severity of the dysmenorrhea (menstrual pain), pelvic pain and dyspareunia (painful sexual intercourse) experienced by participants occurring during the most recent menstrual cycle on a 4-point scale, where 0 = absent, 1 = mild, 2 = moderate, and 3 = severe. Total score was calculated as a sum of the individual pain scores for dysmenorrhea, dyspareunia and pelvic pain. The total score range: 0 (no pain) to 9 (worst possible pain).
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 12 | 14
units on a scale
  Baseline | 7.08 (1.379) | 7.00 (1.109)
  Week 4: number analyzed (Participants) | 9 | 12
  Week 4 | 5.00 (1.871) | 4.58 (2.712)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 2.89 (2.571) | 3.83 (2.443)
  Week 12: number analyzed (Participants) | 12 | 8
  Week 12 | 3.42 (2.575) | 2.63 (1.996)
  Week 16: number analyzed (Participants) | 12 | 12
  Week 16 | 4.83 (3.070) | 3.17 (2.791)

10. Secondary Outcome: Endometriosis Health Profile 30 (EHP-30) Score at Baseline and Week 8
Description: EHP-30 is a validated quality of life (QoL) scale assessing emotional, physical and sexual function. EHP-30 consists of 30 items that assess the frequency of physical and mental manifestations of endometriosis during the previous 4 weeks on a 5-point Likert scale (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always).. Scores for 6 domains (pain, control and powerlessness, emotional well-being, social support, self image, and sexual intercourse) were obtained as a sum of all relevant item scores and transformed to a 0 to 100 score range. Each domain score ranges from 0 (best possible health status) to 100 (worst possible health status).
Time Frame: Baseline and Week 8
Population: Restricted FAS. Here 'number analyzed' signifies those participants who were evaluable for specified category for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale
  Baseline: Pain | 58.97 (14.661) | 56.68 (13.213)
  Baseline: Control & Powerlessness | 69.96 (20.250) | 64.84 (22.098)
  Baseline: Emotional well-being | 52.85 (18.005) | 41.15 (21.671)
  Baseline: Social support | 57.57 (24.701) | 46.48 (26.018)
  Baseline: Self-image | 53.51 (29.700) | 45.31 (27.550)
  Baseline: Sexual intercourse: number analyzed (Participants) | 14 | 14
  Baseline: Sexual intercourse | 58.93 (37.835) | 65.36 (23.490)
  Week 8: Pain: number analyzed (Participants) | 17 | 14
  Week 8: Pain | 28.34 (17.179) | 26.30 (23.325)
  Week 8: Control & Powerlessness: number analyzed (Participants) | 17 | 14
  Week 8: Control & Powerlessness | 28.92 (20.437) | 27.98 (34.298)
  Week 8: Emotional well-being: number analyzed (Participants) | 17 | 14
  Week 8: Emotional well-being | 27.94 (17.664) | 16.37 (19.300)
  Week 8: Social support: number analyzed (Participants) | 16 | 14
  Week 8: Social support | 36.33 (28.706) | 26.34 (30.636)
  Week 8: Self-image: number analyzed (Participants) | 17 | 14
  Week 8: Self-image | 31.86 (23.613) | 24.40 (27.632)
  Week 8: Sexual intercourse: number analyzed (Participants) | 11 | 11
  Week 8: Sexual intercourse | 45.45 (32.822) | 29.20 (31.654)

11. Secondary Outcome: Global Response Assessment (GRA) at Week 8
Description: GRA questionnaire is a 7-point symmetric scale which measures participant-reported overall response to treatment compared to baseline as 1 of the following possible responses: markedly worse, moderately worse, slightly worse, no change, slightly improved, moderately improved, and markedly improved. Number of participants with each response is reported.
Time Frame: Week 8
Population: Restricted FAS. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 17 | 14
Participants
  Markedly Worse | 0 | 1
  Moderately Worse | 0 | 0
  Slightly Worse | 0 | 0
  No Change | 3 | 2
  Slightly Improved | 4 | 2
  Moderately Improved | 8 | 6
  Markedly Improved | 2 | 3

12. Secondary Outcome: Participant Global Satisfaction at Week 8
Description: Participant global satisfaction is assessed using Patient Reported Treatment Impact (PRTI) which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant's response is rated on a 5-point scale where 1 = extremely satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied and 5 = extremely dissatisfied. Number of participants with each response is reported.
Time Frame: Week 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 17 | 14
Participants
  Extremely satisfied | 5 | 3
  Satisfied | 7 | 7
  Neither satisfied nor dissatisfied | 5 | 2
  Dissatisfied | 0 | 0
  Extremely dissatisfied | 0 | 2

13. Secondary Outcome: Participant Global Preference at Week 8
Description: Participant global preference is assessed using PRTI, which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant reported previous treatment under following categories: hormonal contraceptive, painkiller, and hormone treatment by injection, hormone treatment by tablet, surgery, and no treatment. Participant preference was assessed using following categories: definitely prefer study medication, slightly prefer study medication, no preference, slightly prefer previous treatment, and definitely prefer previous treatment. Number of participants under each of the categories is reported. For previous treatment, a single participant may be represented in more than 1 category.
Time Frame: Week 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 17 | 14
Participants
  Hormonal contraceptive | 7 | 7
  Painkiller | 11 | 7
  Hormone treatment by injection | 1 | 1
  Hormone treatment by tablet | 1 | 0
  Surgery | 5 | 5
  No treatment | 4 | 1
  Definitely prefer study medication | 11 | 6
  Slightly prefer study medication | 3 | 3
  No preference | 0 | 2
  Slightly prefer previous treatment | 1 | 1
  Definitely prefer previous treatment | 2 | 2

14. Secondary Outcome: Participant Willingness to Re-use Study Medication
Description: Participant willingness to re-use study medication is assessed using PRTI, which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant willingness to re-use study medication was assessed using following categories: definitely want to re-use, might want to re-use, not sure, might not want to re-use, definitely would not want to re-use.
Time Frame: Week 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 17 | 14
Participants
  Definitely want to re-use | 13 | 7
  Might want to re-use | 1 | 1
  Not sure | 2 | 3
  Might not want to re-use | 1 | 1
  Definitely would not want to re-use | 0 | 2

15. Secondary Outcome: Plasma Nerve Growth Factor (NGF) Concentration
Time Frame: Day 1, Week 8, and Week 16 (End of Treatment)
Population: FAS. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 21 | 24
picogram per milliliter (pg/mL)
  Day 1 | 301 (1217) | 32.7 (10.6)
  Week 8: number analyzed (Participants) | 20 | 20
  Week 8 | 4053 (1276) | 30.7 (7.8)
  Week 16: number analyzed (Participants) | 21 | 20
  Week 16 | 3010 (921) | 31.4 (10.6)

16. Secondary Outcome: Amount of Rescue Medication Used
Description: Mean amount of daily rescue medication (acetaminophen 500 mg tablet/capsule) taken for endometriosis associated pain (in mg) was assessed.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 18 | 15
mg/day
  Baseline | 66.78 (34.60) | 56.60 (61.39)
  Week 4: number analyzed (Participants) | 18 | 14
  Week 4 | 41.78 (38.69) | 48.86 (50.57)
  Week 8: number analyzed (Participants) | 15 | 10
  Week 8 | 34.73 (37.21) | 43.20 (28.95)
  Week 12: number analyzed (Participants) | 16 | 12
  Week 12 | 21.25 (20.57) | 29.33 (28.09)
  Week 16: number analyzed (Participants) | 15 | 10
  Week 16 | 24.13 (27.33) | 28.40 (25.81)

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 113 days after last dose that were absent before treatment or worsened relative to pre-treatment state.
Time Frame: Baseline up to 113 days after last dose of study medication
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 22 | 25
Participants
  AEs | 16 | 21
  SAEs | 0 | 3

18. Secondary Outcome: Number of Participants With New or Worsened Neurological Examinations
Description: A neurological evaluation was performed by a consulting neurologist if adverse events suggested new or worsening peripheral neuropathy with respect to baseline or any adverse event of abnormal peripheral sensation was recorded. A neurological evaluation was done as soon as the above signs and symptoms were known, preferably within 7 days of becoming aware of such problems if possible. Neurological evaluation was done using Neuropathy Impairment Score (NIS) by investigator. Neurologic examination assessment included strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes. Abnormality was judged by the investigator.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each treatment arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 22 | 23
Participants
  Week 2 | 3 | 1
  Week 4: number analyzed (Participants) | 20 | 22
  Week 4 | 0 | 0
  Week 8: number analyzed (Participants) | 20 | 21
  Week 8 | 1 | 1
  Week 12: number analyzed (Participants) | 20 | 19
  Week 12 | 1 | 2
  Week 16: number analyzed (Participants) | 21 | 20
  Week 16 | 1 | 0

19. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Serum samples were analyzed for the presence or absence of anti-tanezumab antibodies using validated semi-quantitative enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 1 (pre-dose), Weeks 2, 4, 8, and 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here 'number analyzed' signifies those participants who were evaluable at specified time point. Only participants who received tanezumab were planned to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 22
Participants
  Day 1: number analyzed (Participants) | 21
  Day 1 | 0
  Week 2 | 0
  Week 4: number analyzed (Participants) | 21
  Week 4 | 0
  Week 8: number analyzed (Participants) | 20
  Week 8 | 0
  Week 16: number analyzed (Participants) | 20
  Week 16 | 0

20. Secondary Outcome: Number of Participants With Positive Urine or Serum Pregnancy Test
Time Frame: Screening, Weeks 2, 4, 8, 12, and Early termination
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 22 | 23
Participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tanezumab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 3/25
Other Adverse Events (participants affected / at risk) | 16/22 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=22) | Placebo (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=22) | Placebo (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Gaze palsy (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Feeling cold (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 2
Temperature intolerance (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 3
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Venomous sting (Injury, poisoning and procedural complications) | 1 | 0
Blood iron decreased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Allodynia (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Facial neuralgia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 4
Hyperreflexia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2
Mental impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 5 | 3
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Peripheral coldness (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Nerve growth factor (NGF) results were reported only for plasma since a reliable assay was not available for analyzing NGF in urine. Study was prematurely terminated and recruitment was stopped due to futility shown in pre-planned interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.